CLINICAL TRIAL: NCT06768450
Title: Online Mindfulness Meditation for Mild Cognitive Impairment and Mild Dementia: a Feasibility Study
Brief Title: Online Meditation for Mild Cognitive Impairment and Mild Dementia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 341708; 341708 (Registry Identifier: The Integrated Research Application System (IRAS) in UK)
Record Dates: First submitted 2024-09-13; First posted 2025-01-10 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2024-09

CONDITIONS: Mild Cognitive Impairment (MCI); Dementia
Keywords: Dementia; Mild cognitive impairment; Feasibility; Acceptability; Online; Mindfulness; Meditation
MeSH Terms: conditions — Cognitive Dysfunction; Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Online mindfulness meditation arm (Experimental): Participants over 60 years old with mild cognitive impairment or mild dementia will be recruited. An 8-week online meditation training program will be provided.
  Interventions: Behavioral: Online mindfulness meditation

INTERVENTIONS:
Behavioral: Online mindfulness meditation — The mindfulness meditation program is adapted from the Breathwork Mindfulness for Stress program. However, it uses shorter meditations designed for individuals who cannot sit for 40 minutes. The mindfulness meditation program encourages greater self-acceptance, kindness, and compassion toward oneself. It builds on this concept by helping participants find pleasure in life despite suffering, fostering kindness and compassion toward others, and increasing social connections to counteract the social isolation common among individuals with chronic and long-term illnesses.
  The program will be led by a well-trained Breathwork mindfulness instructor and conducted remotely via Microsoft Teams once a week for 8 weeks. Each session will last 2 to 2.5 hours and consist of body scans, mindful movements, and various meditations, introducing new ideas every week.

SUMMARY:
The study will look at whether online mindfulness meditation (OMM) is easy for older adults with mild cognitive impairment (MCI) and mild dementia to use. It will also see how OMM affects their mood, sleep, and quality of life.

The investigators will recruit 32 participants, divided into 4 groups of 8 people each.

Participants will:

* Attend an online mindfulness meditation class once a week for 8 weeks
* Practice at home for 20 minutes each day
* Keep a simple record of their practice and feelings

DETAILED DESCRIPTION:
This research aims to investigate the feasibility and acceptability of online meditation for older adults with mild cognitive impairment (MCI) and mild dementia in the UK and to explore its impact on cognitive function, mood, mindfulness, and quality of life. This study will recruit 32 participants with MCI and mild dementia. Participants will receive mindfulness meditation training in an online group-based format, with 8 participants per group in 4 waves. A qualified meditation teacher will lead the sessions via Microsoft Teams once a week for 8 weeks (lasting 2 to 2.5 hours per session).

The study outcomes will include feasibility of the intervention, acceptability to participants, cognitive function, mindfulness, and quality of life. Data will be collected at baseline and after the intervention. A paired t-test will compare pre- and post-intervention changes if the data meet assumptions of normal distribution and homogeneity of variance. Otherwise, non-parametric statistical analyses will be applied.

ELIGIBILITY:
Inclusion Criteria:

* Age 60 years or older.
* MCI: Concern regarding a change in cognition, with impairment in one or more cognitive domains, including memory, executive function, attention, language, and visuospatial skills. Preservation of independence in functional abilities and does not meet the criteria for dementia, as described in the National Institute on Aging and Alzheimer's Association (NIA-AA) diagnostic guidelines.
* Mild dementia: As described in the NIA-AA research framework, mild dementia is defined as substantial progressive cognitive impairment affecting several domains and/or neurobehavioral disturbances. Documented by the individual's report, an observer (e.g., a study partner) report, or by changes observed on longitudinal cognitive testing. Clearly evident functional impact on daily life, mainly affecting instrumental activities. No longer fully independent and requires occasional assistance with daily activities.
* Access to an electronic device (e.g., smartphone, computer, or tablet) and the internet.
* Ability and willingness to provide informed consent by signing the Consent Form.

Exclusion Criteria:

* Current active or past significant experience with meditation.
* Clinically significant mental or physical health disorder beyond MCI or dementia that may affect cognition and/or the ability to complete the study (e.g., severe depression, suicidality, psychosis, post-traumatic stress disorder (PTSD), major psychiatric diagnoses, social anxiety (e.g., difficulty participating in a group setting), or severe impairments in eyesight, hearing, or upper limb motor movements).
* Inability to commit to attending classes (e.g., planning to miss three or more classes).
* Lack of proficiency in English.
* Diagnosed with moderate or severe dementia.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Conversion rate | through study completion, an average of 1 year
  Conversion Rate= Number of participants enrolled / Number of potential participants contacted × 100%
Retention rate | through study completion, an average of 1 year
  Retention Rate (%)= Number of participants who completed the study / Number of participants initially enrolled × 100%
Attrition rate | through study completion, an average of 1 year
  Attrition Rate (%)= Number of participants who dropped out / Total number of participants initially enrolled × 100%
Client Satisfaction Questionnaire | immediately after the intervention
  It is a standardized 8-item tool that has demonstrated good reliability and validity in mental health services. Items are scored from 1 (low satisfaction) to 4 (high satisfaction) with different descriptors for each response point. Total scores range from 8 to 32, with higher scores indicating greater satisfaction.

SECONDARY OUTCOMES:
Modified Telephone Interview for Cognitive Status | baseline and immediately after the intervention
  The Modified Telephone Interview for Cognitive Status is a brief, 13-item test of cognitive functioning with total scores ranging from 0 to 50. Questions of orientation, repetition, naming, and calculations are some of the items covered. Additionally, a 10-item non-semantically related word list is recalled both immediately and after a delay of about 5 minutes filled with distractor questions. Higher scores mean a better outcome.
Pittsburgh sleep quality index | baseline and immediately after the intervention
  It is a self-rated questionnaire which assesses sleep quality and disturbances over a 1-month time interval. Nineteen individual items generate seven component scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. The total scores range from 0 to 21. Higher scores mean a worse outcome.
Hospital anxiety and depression scale | baseline and immediately after the intervention
  It is used in the setting of a general medical hospital outpatient clinic to assess the mental health of patients. It has two subscales (anxiety and depression), each with seven items and a score of 0-3 for each item, the total score is 21 respectively. Higher scores indicate a worse condition.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] You J, Khan Z, Swaroop R, Sun Y, Velayudhan L, Aarsland D. Online mindfulness meditation for mild cognitive impairment and mild dementia: A feasibility study protocol. PLoS One. 2025 Nov 25;20(11):e0336583. doi: 10.1371/journal.pone.0336583. eCollection 2025. PMID 41289241